CLINICAL TRIAL: NCT06942429
Title: Stepped Versus Stratified Care for Anxiety Disorders in Youth: A Pragmatic Non-Inferiority Randomized Controlled Trial
Brief Title: Stepped Versus Stratified Care for Anxiety Disorders in Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Matti Cervin, Associate Professor, Senior Clinical Psychologist, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dnr 2025-01014-01
Record Dates: First submitted 2025-04-09; First posted 2025-04-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Social Anxiety Disorder; Separation Anxiety Disorder; Specific Phobia; Panic Disorder; Generalized Anxiety Disorder; Agoraphobia
Keywords: anxiety disorders; children; adolescents; cognitive behavioral therapy; non-inferiority; care models; stepped care; stratified care
MeSH Terms: conditions — Phobia, Social; Anxiety, Separation; Phobia, Specific; Panic Disorder; Generalized Anxiety Disorder; Agoraphobia; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistical analyst
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stepped Care (Experimental): All participants in stepped care will receive internet-delivered cognitive-behavioral therapy (ICBT) in the first Treatment course (A). Participants who have not responded to treatment or continue to exhibit clinical levels of anxiety severity will be offered personalized in-person CBT in the second Treatment course (B).
  Interventions: Behavioral: Internet-delivered cognitive-behavioral therapy; Behavioral: Personalized in-person cognitive-behavioral therapy
- Stratified Care (Active Comparator): In stratified care, Treatment course A aims to allocate approximately half of the participants to internet-delivered cognitive-behavioral therapy (ICBT) and the other half to personalized in-person CBT, based on their algorithm-generated clinical complexity score. Identical to stepped care, those who have not responded to treatment or continue to exhibit clinical levels of anxiety severity after Treatment course A will be offered personalized in-person CBT in Treatment course B.
  Interventions: Behavioral: Internet-delivered cognitive-behavioral therapy; Behavioral: Personalized in-person cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Internet-delivered cognitive-behavioral therapy — Internet-delivered cognitive behavioral therapy (ICBT) is a 12-module intervention delivered over a maximum of 14 weeks. Two age-specific versions are available: [1] for children aged 8-12 years and [2] for adolescents aged 13-17 years. Both versions share the same core content, but the texts, illustrations, videos, and exercises are adapted to be developmentally appropriate. Each version focuses on exposure, along with psychoeducation, coping strategies, and relapse prevention. Caregivers have access to a parallel program that mirrors the structure of the youth program. Both patients and caregivers engage with a therapist through a secure digital platform, communicating via text messages similar to emails. Two scheduled telephone or videoconference calls are conducted approximately 3-4 and 7-8 weeks into treatment, respectively, to follow up on adherence and address questions related to the intervention. Additional telephone support will be available on demand.
Behavioral: Personalized in-person cognitive-behavioral therapy — Personalized in-person cognitive-behavioral therapy (CBT) follows a manual drawing on previously published protocols and meta-analyses on effective components of CBT for pediatric anxiety disorders and results from our pilot study. It consists of 12 weekly one-hour sessions delivered over a maximum of 14 weeks. It follows a disorder-specific CBT approach, with a strong emphasis on therapist-led exposure tailored to the patient's principal anxiety disorder. Participants receive workbooks containing information on anxiety disorders, the treatment rationale, and the rationale for exposure therapy. The intervention has three phases: [1] 1-2 sessions of psychoeducation and symptom identification, [2] 8-10 sessions of therapist-led exposure with homework, and [3] 1-2 sessions of relapse prevention planning. Caregiver involvement is tailored to the individual needs of each participant, with a maximum of 2 additional hours allocated for caregivers beyond the standard treatment time.

SUMMARY:
The goal of this clinical trial is to compare stepped care to stratified care as overall healthcare models for children and adolescents aged 8-17 with anxiety disorders. It addresses one main question:

• Is stepped care non-inferior to stratified care in supporting participants to achieve a treatment response?

Researchers will compare two care models:

* Stepped care, where all participants begin with 14 weeks of internet-delivered cognitive behavioral therapy (ICBT) and receive an additional 14 weeks of personalized in-person CBT if needed.
* Stratified care, where participants are assigned to either 14 weeks of ICBT or 14 weeks of in-person CBT based on clinical complexity, and may also receive additional 14 weeks of in-person CBT if necessary.

Participants will:

* Be randomly assigned to one of the two care models.
* Complete a wide range of assessments at baseline, during treatment, and at 4, 8, 12, and 24 months, with the 8-month point as the primary endpoint.
* Receive either ICBT, in-person CBT, or both, depending on their care model and response to treatment.
* Participate in ancillary studies involving DNA sampling, cognitive testing, and national registry linkages to help predict treatment response and long-term outcomes.

DETAILED DESCRIPTION:
A detailed description is available in the full study protocol. All study protocol versions can be accessed at the Open Science Framework (https://osf.io/a9qhw/).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 8.0 to 17.5 years. Confirmed by the child and/or caregiver.
2. Principal DSM-5-TR anxiety disorder of social anxiety disorder, generalized anxiety disorder, panic disorder, separation anxiety disorder, specific phobia, or agoraphobia. Confirmed by the structured diagnostic interview (DIAMOND-KID). "Principal" indicates that the anxiety disorder is judged by the clinician to be in most urgent need of treatment (among potential co-occurring disorders).
3. Available caregiver who can support the child in treatment. Confirmed by the caregiver.
4. Child and at least one caregiver can read, write, and communicate in Swedish. Confirmed by the child and/or caregiver.
5. Child (≥13 years) and caregiver have access to a Swedish electronic identification (BankID or Freja eID).
6. Access to the internet. Confirmed by the child and/or caregiver.
7. Ability to attend in-person CBT sessions at the clinic. Confirmed by the child and/or caregiver.

Exclusion Criteria:

1. Principal DSM-5-TR anxiety disorder of specific phobia concerning the domain of blood-injection-injury (due to the ICBT program not including relevant information on applied-tension techniques to avoid fainting during exposure exercises). Confirmed by a specific phobia of this sort being classified as the most functionally impairing anxiety disorder during the structured diagnostic interview (DIAMOND-KID).
2. Ongoing psychological treatment for an anxiety disorder. Confirmed by the child and/or caregiver.
3. Social/familial/educational difficulties in more immediate need of management than an anxiety disorder. Confirmed by the assessor through information from the child and/or caregiver and/or other available sources.
4. Immediate risk to self or others that require urgent attention, such as suicidality. Confirmed by the assessor through information from the child and/or caregiver and other available sources.
5. The potential participant has a relative (e.g., sibling, cousin) included in the study. Confirmed by the assessor through information from the caregiver and other available sources.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 556 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2029-11-05 (Estimated); Study Completion 2031-03-05 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impressions - Improvement Scale | 4 months (17-20 weeks post-randomization); 8 months (35-40 weeks post-randomization, primary endpoint); 12 months (53-60 weeks post-randomization, observational follow-up); 24 months (105-116 weeks post-randomization, observational follow-up)
  The Clinical Global Impressions - Improvement (CGI-I) Scale is a 1-item measure where a trained interviewer uses all available information about the patient to rate improvement on a 7-point scale: 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse. In this study, improvement on the CGI-I is assessed by comparing the current status of the participant to their baseline condition. In line with previous studies, a score of 1 or 2 on the CGI-I is classified as a treatment response and scores of 3 to 7 as non-response. This binary variable is the primary outcome of the trial.

SECONDARY OUTCOMES:
Pediatric Anxiety Rating Scale | Baseline; 4 months (17-20 weeks post-randomization); 8 months (35-40 weeks post-randomization, primary endpoint); 12 months (53-60 weeks post-randomization, observational follow-up); 24 months (105-116 weeks post-randomization, observational follow-up)
  The Pediatric Anxiety Rating Scale (PARS) is a clinician-rated measure of overall anxiety severity. It includes seven items assessing the number of anxiety symptoms, their frequency, anxiety-related avoidance, anxiety-related distress, physical symptoms of anxiety, family interference, and social interference. In the current study, in accordance with other trials for youth anxiety disorders, the 6-item version of PARS is used which excludes the item assessing number of symptoms. The resulting 6-item scale yields a score of 0 to 30, with higher scores indicating more severe anxiety.
Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders - Child and Adolescent Version | Baseline; 4 months (17-20 weeks post-randomization); 8 months (35-40 weeks post-randomization, primary endpoint); 12 months (53-60 weeks post-randomization, observational follow-up); 24 months (105-116 weeks post-randomization, observational follow-up)
  The Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders - Child and Adolescent Version (DIAMOND-KID) is a semi-structured interview that assesses the most common mental disorders in children and adolescents, including all the anxiety disorders used for inclusion in the present study. The full interview is conducted at baseline and at the 12- and 24-month post-randomization assessments. A shortened version that includes anxiety disorders and major depression is conducted at the 4- and 8-month post-randomization assessments. Data from the DIAMOND-KID will be used to evaluate the proportion who no longer meet diagnostic criteria for [1] their principal baseline anxiety disorder and [2] any anxiety disorder.
Clinical Global Impressions Scale-Severity | Baseline; 4 months (17-20 weeks post-randomization); 8 months (35-40 weeks post-randomization, primary endpoint); 12 months (53-60 weeks post-randomization, observational follow-up); 24 months (105-116 weeks post-randomization, observational follow-up)
  The Clinical Global Impressions Scale-Severity (CGI-S) is a single-item measure where a trained assessor makes an overall severity rating of a specific disorder accounting for all available information about the patient, including but not limited to current symptoms, impairment, and general functioning. In this study, in line with previous trials of youth anxiety disorders, the CGI-S is used to rate the overall severity of the patient's anxiety symptoms, irrespective of their association with a specific anxiety disorder.
Children's Global Assessment Scale | Baseline; 4 months (17-20 weeks post-randomization); 8 months (35-40 weeks post-randomization, primary endpoint); 12 months (53-60 weeks post-randomization, observational follow-up); 24 months (105-116 weeks post-randomization, observational follow-up)
  The Children's Global Assessment Scale (CGAS) is a clinician-rated one-item scale of psychosocial functioning/impairment, ranging from 1 to 100 with higher scores indicating better functioning.
Revised Children's Anxiety and Depression Scale | Baseline; 4 months (17-20 weeks post-randomization); 8 months (35-40 weeks post-randomization, primary endpoint); 12 months (53-60 weeks post-randomization, observational follow-up); 24 months (105-116 weeks post-randomization, observational follow-up)
  The Revised Children's Anxiety and Depression Scale (RCADS) is a patient- and caregiver-reported questionnaire assessing specific anxiety symptoms and their frequency. The original version includes 47 items. In the present study, we use the 30-item version, which maintains the factor structure of the original version and demonstrates conserved psychometric properties. The RCADS has shown adequate psychometric properties in several studies, including in Swedish youth, and is an internationally recommended measure for the assessment of internalizing symptoms in children and adolescents. Both patient- and caregiver-reported versions are used in the study. We will use the subscale that sums all the anxiety symptoms, which ranges from 0 to 60, with higher scores indicating more frequent anxiety symptoms.
Child Anxiety Life Interference Scale-Revised | Baseline; 4 months (17 to 20 weeks post-randomization); 8 months (35 to 40 weeks post-randomization, primary endpoint); 12 months; 24 months
  The Child Anxiety Life Interference Scale-Revised (CALIS-R) is a patient- and caregiver-reported measure of interference associated with youth anxiety. The measure is an internationally recommended tool for the assessment of interference stemming from anxiety in children and adolescents. The patient-reported version consists of 9 items, each rated on a 0-4 response scale, resulting in a total score of 0 to 36, with higher overall scores indicating more interference. The caregiver-reported version consists of two sub-scales, where one sub-scale assesses interference for the child (9 items; range: 0 to 36) and the other interference for the family (8 items; range: 0 to 32), with higher scores indicating more interference. For the caregiver-reported version, the two sub-scales will be reported separately.
Proportion of participants who do not adhere to the assigned treatment/s | 4 months (17-20 weeks post-randomization); 8 months (35-40 weeks post-randomization, primary endpoint)
  Non-adherence to treatment is defined as completing fewer than six modules of ICBT, attending fewer than six sessions of personalized in-person CBT, or discontinuing/refusing treatment despite clinical judgment indicating it is warranted. An exception to the six-module/session rule is made if treatment is discontinued due to substantial symptom improvement to non-clinical levels, with therapist agreement that further treatment is unnecessary. At 4 months, non-adherence is assessed based on the first course of treatment. At 8 months, it is assessed based on overall adherence across both treatment courses: [0] complete adherence (adhering to all assigned treatments), [1] partial adherence (adhering to one but not all assigned treatments), or [2] full non-adherence (adhering to no assigned treatment).
Adverse events | 4 months (17-20 weeks post-randomization); 8 months (35-40 weeks post-randomization, primary endpoint)
  Adverse events are continuously screened, recorded, and monitored by study personnel and through the patient- and caregiver-reported Adverse Events Questionnaire, which includes 22 predefined events and an open-ended option. Events will be reported as the total number of documented events, ranging from 0 with no defined upper limit.

OTHER OUTCOMES:
Health economic outcomes | Baseline; 4 months (17-20 weeks post-randomization); 8 months (35-40 weeks post-randomization, primary endpoint); 12 months (53-60 weeks post-randomization, observational follow-up); 24 months (105-116 weeks post-randomization, observational follow-up)
  Health economic evaluations, including the calculation of Incremental Cost-Effectiveness Ratios (ICER) and assessment of willingness-to-accept thresholds, will be performed. The details will be specified in a separate Health Economic Analysis Plan (HEAP) and the planned approach is available in the full study protocol at Open Science Framework (https://osf.io/a9qhw/). These measures will not be used to make inference about the non-inferiority RCT regarding anxiety outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Matti Cervin, PhD, Principal Investigator — Lund University & CAMHS Skåne; Eva Serlachius, MD, PhD, Principal Investigator — Lund University & CAMHS Skåne
Locations (1):
- Forskningsmottagning Barn och ungdomspsykiatri Lund, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
The data are pseudonymized according to national (Swedish) and European Union legislation and cannot be anonymized and published in an open repository. Participants in the study consent for their data to be shared with other international researchers for research purposes. The data can be made available upon reasonable request on a case-by-case basis according to the current legislation and ethical permits.

REFERENCES:
- See also: All versions of the study protocol are shared on the Open Science Framework platform. The trial includes an ancillary study, fully described in the study protocol, designed to identify predictive markers of treatment response and long-term outcomes. — https://osf.io/a9qhw/